CLINICAL TRIAL: NCT02646423
Title: Effect of a Patient-Centered Decision App on TOLAC: An RCT
Brief Title: Effect of a Patient-Centered Decision App on TOLAC
Acronym: PROCEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Northwestern Memorial Hospital (Other); Massachusetts General Hospital (Other); Marin Community Clinics (Other); Sutter Health (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01HD078748 (NIH); 1R01HD078748 (NIH)
Record Dates: First submitted 2015-12-15; First posted 2016-01-05 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Pregnancy; Repeat Cesarean Section; Vaginal Births After Cesarean
Keywords: Trial of labor after cesarean; Elective repeat cesarean delivery; Decision tool; Shared decision making

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prior CD Decision App (PCDDA) (Experimental): Women who are randomized to PCDDA will be provided access to a tablet which they can use to view the Prior CD Decision App at their own pace. The research assistant will print a summary of the participant's predicted likelihood of a vaginal delivery (VBAC) if she undergoes a trial of labor (TOLAC), as well as her answers to the values clarification exercises, that she can review and share with whomever she chooses, including her provider.
  Interventions: Behavioral: Prior CD Decision App
- Usual Care - No App (No Intervention): Women randomized to the Usual Care - No App group will simply continue with usual care.

INTERVENTIONS:
Behavioral: Prior CD Decision App — The Prior CD Decision App begins with an explanation that its goal is to help the user better understand the two approaches to delivery she is eligible for (trial of labor after cesarean (TOLAC) and elective repeat cesarean delivery (ERCD)), and that its goal is to help her engage with her provide in making an informed, shared decision regarding which approach to undergo. It includes four sections: a calculator to estimate the likelihood of having a vaginal delivery if she undergoes TOLAC, a series of information pages that include graphical presentations of the chances of various potential outcomes of the two options, a series of values clarification exercises to help the user think through what's important to her, and a summary print out for her to keep.
  Arms: Prior CD Decision App (PCDDA)

SUMMARY:
Cesarean delivery (CD) is the most common inpatient surgery in the US, accounting for nearly one third of births annually. In the last decade, the CD rate has increased by approximately 50%, with almost 1.3 million procedures performed in 2012 (Hamilton 2013). CDs have been associated with an increase in major maternal morbidity (Silver 2010), with corresponding increases in length of inpatient care following delivery and frequency of hospital readmission (Lydon-Rochelle 2000). Organizations including Healthy People, the American College of Obstetricians and Gynecologists (ACOG), and the American College of Nurse Midwives have targeted reducing the CD rate as an important public health goal for more than a decade; however, identifying interventions to achieve this goal has proven challenging.

Repeat CDs are a significant contributor to the increased cesarean rate, resulting from the combination of a rising rate of primary CD and a decreasing rate of vaginal birth after cesarean (VBAC), which declined from a high of 28.3% in 1996 (Guide 2010) to 9.2% in 2010 (Hamilton 2011). Why the VBAC rate has decreased so dramatically remains a subject of debate; the extent to which these changes are driven by patient preferences is not known. An NIH consensus conference statement noted that "the informed consent process for TOLAC and Elective Repeat Cesarean Delivery (ERCD) should be evidence-based, minimize bias, and incorporate a strong emphasis on the values and preferences of pregnant women," and recommended "interprofessional collaboration to refine, validate, and implement decision-making and risk assessment tools" to accomplish that goal (Cunningham 2010).

Our group recently created a decision tool, which we refer to as the Prior CD App (PCDA), to help English- or Spanish-speaking TOLAC-eligible women delivering at hospitals that offer TOLAC consider individualized risk assessments, incorporate their values and preferences, and participate in a shared decision making process with their providers to make informed decisions about delivery approach. We are now conducting a randomized study of the effect of a Prior CD App on TOLAC and VBAC rates, as well as a number of aspects of decision quality.

ELIGIBILITY:
Inclusion Criteria:

1. Women with exactly one prior Cesarean Delivery.
2. Current singleton pregnancy.
3. Gestational age, 12-24 weeks.
4. English or Spanish speaker.
5. Must be receiving prenatal care at one of the participating centers.

Exclusion Criteria:

1. Contraindications to vaginal delivery (e.g., placenta previa, prior classical cesarean, previous uterine rupture).
2. Prior VBAC.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1485 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Kupperman, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (5):
- United States (5):
  - Sutter Health, California Pacific Medical Center, St. Luke's Campus, San Francisco, California
  - UCSF, San Francisco, California
  - Marin Community Clinic, San Rafael, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Bernstein SN, Matalon-Grazi S, Rosenn BM. Trial of labor versus repeat cesarean: are patients making an informed decision? Am J Obstet Gynecol. 2012 Sep;207(3):204.e1-6. doi: 10.1016/j.ajog.2012.06.057. Epub 2012 Jul 4. PMID 22939727
- [Background] Farnworth A, Robson SC, Thomson RG, Watson DB, Murtagh MJ. Decision support for women choosing mode of delivery after a previous caesarean section: a developmental study. Patient Educ Couns. 2008 Apr;71(1):116-24. doi: 10.1016/j.pec.2007.11.020. Epub 2008 Feb 6. PMID 18255248
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294
- [Background] Kriston L, Scholl I, Holzel L, Simon D, Loh A, Harter M. The 9-item Shared Decision Making Questionnaire (SDM-Q-9). Development and psychometric properties in a primary care sample. Patient Educ Couns. 2010 Jul;80(1):94-9. doi: 10.1016/j.pec.2009.09.034. Epub 2009 Oct 30. PMID 19879711
- [Background] Holmes-Rovner M, Kroll J, Schmitt N, Rovner DR, Breer ML, Rothert ML, Padonu G, Talarczyk G. Patient satisfaction with health care decisions: the satisfaction with decision scale. Med Decis Making. 1996 Jan-Mar;16(1):58-64. doi: 10.1177/0272989X9601600114. PMID 8717600
- [Background] Hamilton BE, Martin JA, Ventura SJ. Births: preliminary data for 2012. Natl Vital Stat Rep. 2013 Sep;62(3):1-20. PMID 24321416
- [Background] Guise J-M, Eden K, Emeis C, Denman MA, Marshall N, Fu R, Janik R, Nygren P, Walker M, McDonagh M. Vaginal birth after cesarean: New insights. Evidence report/Technology assessment no.191. (prepared by the Oregon Health & Science University Evidence-based Practice Center under contract no. 290-2007-10057-I). AHRQ publication no. 10-E003. Rockville, MD: Agency for Healthcare Research and Quality. March 2010.
- [Background] Martin JA, Hamilton BE, Ventura SJ, Osterman MJ, Kirmeyer S, Mathews TJ, Wilson EC. Births: final data for 2009. Natl Vital Stat Rep. 2011 Nov 3;60(1):1-70. PMID 22670489
- [Background] Grobman WA, Lai Y, Landon MB, Spong CY, Rouse DJ, Varner MW, Caritis SN, Harper M, Wapner RJ, Sorokin Y; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. The change in the rate of vaginal birth after caesarean section. Paediatr Perinat Epidemiol. 2011 Jan;25(1):37-43. doi: 10.1111/j.1365-3016.2010.01169.x. Epub 2010 Oct 25. PMID 21133967
- [Background] Landon MB, Hauth JC, Leveno KJ, Spong CY, Leindecker S, Varner MW, Moawad AH, Caritis SN, Harper M, Wapner RJ, Sorokin Y, Miodovnik M, Carpenter M, Peaceman AM, O'Sullivan MJ, Sibai B, Langer O, Thorp JM, Ramin SM, Mercer BM, Gabbe SG; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Maternal and perinatal outcomes associated with a trial of labor after prior cesarean delivery. N Engl J Med. 2004 Dec 16;351(25):2581-9. doi: 10.1056/NEJMoa040405. Epub 2004 Dec 14. PMID 15598960
- [Background] Macones GA, Peipert J, Nelson DB, Odibo A, Stevens EJ, Stamilio DM, Pare E, Elovitz M, Sciscione A, Sammel MD, Ratcliffe SJ. Maternal complications with vaginal birth after cesarean delivery: a multicenter study. Am J Obstet Gynecol. 2005 Nov;193(5):1656-62. doi: 10.1016/j.ajog.2005.04.002. PMID 16260206
- [Background] Lavin JP, Stephens RJ, Miodovnik M, Barden TP. Vaginal delivery in patients with a prior cesarean section. Obstet Gynecol. 1982 Feb;59(2):135-48. PMID 7078857
- [Background] Silver RM. Delivery after previous cesarean: long-term maternal outcomes. Semin Perinatol. 2010 Aug;34(4):258-66. doi: 10.1053/j.semperi.2010.03.006. PMID 20654776
- [Background] Lydon-Rochelle M, Holt VL, Martin DP, Easterling TR. Association between method of delivery and maternal rehospitalization. JAMA. 2000 May 10;283(18):2411-6. doi: 10.1001/jama.283.18.2411. PMID 10815084
- [Result] Kuppermann M, Kaimal AJ, Blat C, Gonzalez J, Thiet MP, Bermingham Y, Altshuler AL, Bryant AS, Bacchetti P, Grobman WA. Effect of a Patient-Centered Decision Support Tool on Rates of Trial of Labor After Previous Cesarean Delivery: The PROCEED Randomized Clinical Trial. JAMA. 2020 Jun 2;323(21):2151-2159. doi: 10.1001/jama.2020.5952. PMID 32484533
- See also: Decisional Conflict Scale — https://decisionaid.ohri.ca/docs/develop/User_Manuals/UM_Decisional_Conflict.pdf
- See also: Decision Self-Efficacy Scale — https://decisionaid.ohri.ca/docs/develop/User_Manuals/UM_Decision_SelfEfficacy.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prior CD Decision App (PCDDA) | Usual Care - No App
Started | 742 | 743
Completed | 735 | 735
Not Completed | 7 | 8
Not completed — Adverse Event | 5 | 7
Not completed — Ineligible | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prior CD Decision App (PCDDA) | Usual Care - No App | Total
Number analyzed (Participants) | 735 | 735 | 1470
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (4.6) | 34.0 (4.5) | 34.0 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 735 | 735 | 1470
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race or ethnic group: White | 394 | 411 | 805
  Race or ethnic group: Latina | 124 | 124 | 248
  Race or ethnic group: Asian or Pacific Islander | 110 | 106 | 216
  Race or ethnic group: Black | 64 | 52 | 116
  Race or ethnic group: Biracial or multiracial/multiethnic | 23 | 25 | 48
  Race or ethnic group: Other | 20 | 17 | 37
Region of Enrollment [Count of Participants; unit: Participants]
  United States: University of California, San Francisco | 192 | 193 | 385
  United States: Marin Community Clinic, San Rafael, California | 26 | 25 | 51
  United States: St Luke's Women's Clinic, San Francisco | 18 | 18 | 36
  United States: Massachusetts General Hospital, Boston | 274 | 278 | 552
  United States: Northwestern University Medical Center, Chicago | 225 | 221 | 446

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Underwent a Trial of Labor After Cesarean (TOLAC) Delivery
Description: Number of participants who underwent a trial of labor after cesarean (TOLAC) delivery, as noted in the medical record.
Time Frame: 0-8 weeks after delivery
Population: Prior CD Decision App (PCDDA): no data available for N=8 participants who delivered at outside institution and no chart or outside questionnaire obtained.
  Usual Care - No App: no data available for N=3 participants who delivered at outside institution and no chart or outside questionnaire obtained.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior CD Decision App (PCDDA) | Usual Care - No App
Number analyzed (Participants) | 727 | 732
Participants | 315 | 338
Statistical Analysis 1: Comparison: Prior CD Decision App (PCDDA) vs Usual Care - No App; Test type: Superiority; Risk Ratio (RR) = 0.94, 95% CI 2-sided [0.84 to 1.05]

2. Secondary Outcome: Number of Participants Who Underwent Vaginal Birth After Cesarean (VBAC)
Description: Number of participants who underwent vaginal birth after cesarean (VBAC), as noted in the medical record.
Time Frame: 0 to 8 weeks after delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Prior CD Decision App (PCDDA) | Usual Care - No App
Number analyzed (Participants) | 727 | 732
Participants | 231 | 233
Statistical Analysis 1: Comparison: Prior CD Decision App (PCDDA) vs Usual Care - No App; Test type: Superiority; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.86 to 1.16]

3. Secondary Outcome: Knowledge About TOLAC and ERCD
Description: 8-item knowledge scale, administered during telephone interview. Scores ranged from 0 to 8 with higher scored indicating greater knowledge.
Time Frame: Approx 34-37 weeks gestation
Population: Prior CD Decision App (PCDDA): 676 Follow-up telephone interviews obtained, 31 Could not be reached for follow-up, 26 Delivered prior to follow-up interview, 2 Had pregnancy loss ≥22 wk.
  Usual Care - No App: 681 Follow-up telephone interviews obtained, 31 Could not be reached for follow-up, 23 Delivered prior to follow-up interview.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior CD Decision App (PCDDA) | Usual Care - No App
Number analyzed (Participants) | 676 | 681
score on a scale | 5.0 (1.8) | 5.0 (1.7)
Statistical Analysis 1: Comparison: Prior CD Decision App (PCDDA) vs Usual Care - No App; Test type: Superiority; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.16 to 0.19]

4. Secondary Outcome: Decisional Conflict
Description: 16-item Decisional Conflict Scale with 5 response categories, administered during telephone interview. Scoring: total scale-0 (no decisional conflict) to 100 (extreme decisional conflict) lower values indicate lower decisional conflict.
Time Frame: Approx 34-37 weeks gestation
Population: Prior CD Decision App (PCDDA): 676 Follow-up telephone interviews obtained. Responses on the Decisional Conflict Scale missing for 5 participants with PCDAA.
  Usual Care-No App: 681 Follow-up interviews obtained. Responses on the Decisional Conflict Scale missing for 6 participants with usual care.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior CD Decision App (PCDDA) | Usual Care - No App
Number analyzed (Participants) | 671 | 675
score on a scale | 17.2 (12.9) | 17.5 (13.9)
Statistical Analysis 1: Comparison: Prior CD Decision App (PCDDA) vs Usual Care - No App; Test type: Superiority; Mean Difference (Net) = -0.38, 95% CI 2-sided [-1.81 to 1.05]

5. Secondary Outcome: Shared Decision Making
Description: 9-item Shared Decision Making Scale, administered during telephone interview.
  Shared decision-making was measured using the 9-item Shared Decision Making Questionnaire (SDM-Q-9), a psychometrically evaluated tool. The core instrument consists of nine statements, which can be rated on a six-point scale from "completely disagree" (0) to "completely agree" (5). The Shared Decision Score can range from 0 to 100, with higher scores indicating more shared decision-making.
Time Frame: Approx 34-37 weeks gestation
Population: Prior CD Decision App (PCDDA): 676 Follow-up telephone interviews obtained. Responses on the Shared Decision Making Scale missing for 12 participants with PCDAA.
  Usual Care-No App: 681 Follow-up interviews obtained. Responses on the Shared Decision Making Scale missing for 9 participants with usual care.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior CD Decision App (PCDDA) | Usual Care - No App
Number analyzed (Participants) | 664 | 672
score on a scale | 74.4 (14.9) | 74.8 (15.9)
Statistical Analysis 1: Comparison: Prior CD Decision App (PCDDA) vs Usual Care - No App; Test type: Superiority; Mean Difference (Net) = -0.34, 95% CI 2-sided [-1.96 to 1.27]

6. Secondary Outcome: Decision Self-Efficacy
Description: 11-item Decisional Self-Efficacy Scale, administered during telephone interview.
  The total score is calculated by summing the 11 items, dividing by 11 and multiplying by 25. Scores range from 0 (not confident) to 100 (extremely confident).
Time Frame: Approx 34-37 weeks gestation
Population: Prior CD Decision App (PCDDA): 676 Follow-up telephone interviews obtained. Responses on the Decisional Self-Efficacy Scale missing for 6 participants with PCDAA.
  Usual Care-No App: 681 Follow-up interviews obtained. Responses on the Decisional Self-Efficacy Scale missing for 9 participants with PCDAA.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior CD Decision App (PCDDA) | Usual Care - No App
Number analyzed (Participants) | 670 | 672
score on a scale | 90.7 (12.3) | 90.3 (12.2)
Statistical Analysis 1: Comparison: Prior CD Decision App (PCDDA) vs Usual Care - No App; Test type: Superiority; Mean Difference (Net) = 0.36, 95% CI 2-sided [-0.94 to 1.66]

7. Secondary Outcome: Decision Satisfaction
Description: 6-item Satisfaction with Decision Scale, administered during telephone interview.
  Satisfaction With Decision Scale scores range from 0 to 5, with higher scores indicating more satisfaction.
Time Frame: Approx 34-37 weeks gestation
Population: Prior CD Decision App (PCDDA): 676 Follow-up telephone interviews obtained. Responses on the Decisional Satisfaction Scale missing for 1 participant with PCDAA.
  Usual Care-No App: 681 Follow-up interviews obtained. Responses on the Decisional Satisfaction Scale missing for 2 participants with PCDAA.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior CD Decision App (PCDDA) | Usual Care - No App
Number analyzed (Participants) | 675 | 679
score on a scale | 4.62 (0.59) | 4.65 (0.54)
Statistical Analysis 1: Comparison: Prior CD Decision App (PCDDA) vs Usual Care - No App; Test type: Superiority; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.09 to 0.03]

8. Secondary Outcome: Maternal Major Morbidity
Description: Defined as any of: uterine rupture, hysterectomy, surgical injury (bowel, bladder/ureter, or other), maternal death, as noted in the medical record for her delivery.
Time Frame: Collected 0 to 8 weeks after delivery.
Population: PCDDA: 15 delivered at outside institution and outcome for maternal major morbidity was not obtained.
  Usual Care- No app: 12 delivered at outside institution and outcome for maternal major morbidity was not obtained.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior CD Decision App (PCDDA) | Usual Care - No App
Number analyzed (Participants) | 720 | 723
Participants | 19 | 23
Statistical Analysis 1: Comparison: Prior CD Decision App (PCDDA) vs Usual Care - No App; Test type: Superiority; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.46 to 1.51]

9. Secondary Outcome: Maternal Minor Morbidity
Description: Defined as any of: blood transfusion, postpartum febrile morbidity (endometritis, cellulitis, urinary tract infection, or other infection), as noted in the medical record for her delivery.
Time Frame: Collected 0 to 8 weeks after delivery.
Population: PCDDA: 15 Delivered at outside institution and maternal minor morbidity outcome not collected during chart review. 1 additional without complete chart review information.
  No App: 12 Delivered at outside institution and maternal minor morbidity outcome not collected during chart review. 1 additional without complete chart review information.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior CD Decision App (PCDDA) | Usual Care - No App
Number analyzed (Participants) | 719 | 722
Participants | 36 | 36
Statistical Analysis 1: Comparison: Prior CD Decision App (PCDDA) vs Usual Care - No App; Test type: Superiority; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.64 to 1.56]

10. Secondary Outcome: 3rd or 4th Degree Lacerations
Description: 3rd or 4th degree lacerations, as noted in the medical record for her delivery.
Time Frame: Collected 0 to 8 weeks after delivery.
Population: PCDDA: 15 delivered at outside institution and outcome for 3rd or 4th degree lacerations was not obtained.
  Usual Care- No app: 12 delivered at outside institution and outcome for 3rd or 4th degree lacerations was not obtained.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior CD Decision App (PCDDA) | Usual Care - No App
Number analyzed (Participants) | 720 | 723
Participants | 16 | 12
Statistical Analysis 1: Comparison: Prior CD Decision App (PCDDA) vs Usual Care - No App; Test type: Superiority; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.64 to 2.81]

11. Secondary Outcome: Perinatal Death or Hypoxic-ischemic Encephalopathy
Description: Stillbirth/fetal demise (antepartum or intrapartum), neonatal death, HIE, as noted in the medical record for her delivery.
Time Frame: Collected 0 to 8 weeks after delivery.
Population: PCDDA: 15 delivered at outside institution and outcome for perinatal death or hypoxic-ischemic encephalopathy was not obtained from chart review.
  No app: 12 delivered at outside institution and outcome for perinatal death or hypoxic-ischemic encephalopathy was not obtained from chart review. 1 delivery at institution missing outcome from chart.
Measure: Number; unit: participants
Arm/Group | Prior CD Decision App (PCDDA) | Usual Care - No App
Number analyzed (Participants) | 720 | 722
participants
  Neonatal death | 2 | 0
  Intrauterine fetal demised | 4 | 0
  Hypoxic-ischemic encephalopathy | 2 | 4
Statistical Analysis 1: Comparison: Prior CD Decision App (PCDDA) vs Usual Care - No App; Test type: Superiority; Risk Ratio (RR) = 2.00, 95% CI 2-sided [0.60 to 6.62]

12. Secondary Outcome: Neonatal Respiratory Morbidity
Description: Respiratory morbidity requiring CPAP or intubation, as noted in the medical record for her delivery.
Time Frame: Collected 0 to 8 weeks after delivery.
Population: PCDDA: 15 delivered at outside institution and neonatal respiratory morbidity was not obtained from chart review. 1 delivery at institution missing outcome from chart.
  No app: 12 delivered at outside institution and neonatal respiratory morbidity was not obtained from chart review. 2 deliveries at institution missing outcome from chart.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior CD Decision App (PCDDA) | Usual Care - No App
Number analyzed (Participants) | 719 | 721
Participants | 67 | 68
Statistical Analysis 1: Comparison: Prior CD Decision App (PCDDA) vs Usual Care - No App; Test type: Superiority; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.72 to 1.35]

13. Secondary Outcome: Neonatal Intensive Care Unit (NICU) Admission
Description: Neonatal intensive care unit (NICU) admission, as noted in the medical record for her delivery.
Time Frame: Collected 0 to 8 weeks after delivery.
Population: Prior CD Decision App (PCDDA): 15 delivered at outside institution and NICU admission was not obtained from chart review.
  Usual Care-No app: 12 delivered at outside institution and NICU admission was not obtained from chart review. 1 delivery at institution missing outcome from chart.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior CD Decision App (PCDDA) | Usual Care - No App
Number analyzed (Participants) | 720 | 722
Participants | 98 | 87
Statistical Analysis 1: Comparison: Prior CD Decision App (PCDDA) vs Usual Care - No App; Test type: Superiority; Risk Ratio (RR) = 1.13, 95% CI 2-sided [0.86 to 1.48]

ADVERSE EVENTS:
Time Frame: Data collection stared on January 2016 and concluded on July 2019. Adverse event data was collected over the entire study time period (3 years, 6 months). Participants were enrolled between 12 to 24 weeks gestation and followed until after delivery. Adverse event data for participants were collected from the date of enrollment until they completed the study at delivery (approximately 1 year).
Description: Prior CD Decision App PCDDA: 7 Did not use decision support tool and/or did not complete study, 8 Delivered at outside institution and no chart or outside questionnaire obtained.
  Usual Care - No App: 8 Did not receive usual care and/or did not complete study, 3 Delivered at outside institution and no chart or outside questionnaire obtained,1 did not have complete chart review information for delivery outcomes, and 1 did not have chart review information for infant morbidity and/or mortality.
Arm/Group | Prior CD Decision App (PCDDA) | Usual Care - No App
All-Cause Mortality (participants affected / at risk) | 0/727 | 0/732
Serious Adverse Events (participants affected / at risk) | 0/727 | 0/732
Other Adverse Events (participants affected / at risk) | 0/727 | 0/732

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT02646423/Prot_SAP_000.pdf